CLINICAL TRIAL: NCT07407023
Title: Randomized Clinical Trial of (PoRI) Post-Stroke Hand Rehabilitation Device
Brief Title: PoRI Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000041770
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Post Stroke; Post Stroke Hand Rehabilitation
Keywords: sensorimotor hand dysfunction

STUDY DESIGN:
Intervention Model Description: The study population only includes patients who present for follow up management of sensorimotor hand dysfunction (muscle strength less than or equal to 3/5) at the Yale New Haven Hospital's Physical Medicine & Rehabilitation (PM&R) department's Inpatient Rehabilitation Unit.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Portable Rehabilitation Interface (PoRI) (Experimental): Participants will receive 20-minute sessions, 3 times per week for 2 to 3 weeks using the PoRI
  Interventions: Device: Portable Rehabilitation Interface (PoRI)
- Standard of care (No Intervention): Participants will receive 20-minute sessions, 3 times per week for 2 to 3 weeks using standard of care

INTERVENTIONS:
Device: Portable Rehabilitation Interface (PoRI) — Handheld device known as the Portable Rehabilitation Interface (PoRI) that moves the hand of patients with sensorimotor hand dysfunction
  Arms: Portable Rehabilitation Interface (PoRI)

SUMMARY:
This randomized clinical trial compares the Portable Rehabilitation Interface (PoRI) device for rehabilitation of hand motor function in post-stroke patients with conventional hand therapy.

ELIGIBILITY:
Inclusion Criteria:

* Between 2 days and a maximum of 2 months have passed since the stroke event
* 0-3/5 muscle strength
* Participants with paralysis or sensorimotor function problems of the fingers of one or both hands.
* Participants must be able to fit their hand comfortably into the device.

Exclusion Criteria:

* Less than 2 days or greater than 2 months have passed since the stroke event
* 4-5/5 muscle strength
* Vulnerable populations.
* Inability of fingers and wrist to stretch to neutral during passive range of motion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) score | Baseline and Week 2-3
  Fugl-Meyer Assessment (FMA) score to assess function with a total score of 100 points. Higher scores mean better recovery, with 0-50 indicating severe impairment and 95-100 showing minimal impairment in motor function, guiding rehabilitation progress.
Box-and-Block Tests (BBT) score | Baseline and Week 2-3
  A Box-and-Block Test (BBT) score is the total number of small blocks a person moves from one section of a divided box to another within 60 seconds. More blocks moved equals greater dexterity.
Visual Analog Scale (VAS) Pain score | Baseline and Week 2-3
  The VAS pain scale is a tool for assessing pain intensity. Participants will be asked to mark a point on a 100 mm horizontal line that represents the intensity of their pain. This line has two endpoints: 0: No pain and 100: Worst possible pain imaginable. The distance from the "0" to the mark is measured in millimeters with the resulting number (0-100) being the VAS pain score
Short Form McGill Pain Questionnaire (sfMPQ) score | Baseline and Week 2-3
  The sfMPQ is scored by summing the values of words that best describe a person's pain. The score ranges from 0 (no pain) to 45 (severe pain).

SECONDARY OUTCOMES:
Device usability and accessibility survey | Week 2-3
  Device usability and accessibility will be evaluated through a patient and researcher survey in the PoRi arm..

CONTACTS AND LOCATIONS:
Overall Officials: Necolle Morgado-Vega, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital's Inpatient Rehabilitation Unit, Milford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No